CLINICAL TRIAL: NCT00494234
Title: A Phase II, Open-label, Non-comparative, International, Multicentre Study to Assess the Efficacy and Safety of KU-0059436 Given Orally Twice Daily in Patients With Advanced BRCA1- or BRCA2-associated Breast Cancer.
Brief Title: Study to Assess The Efficacy and Safety of a PARP Inhibitor For The Treatment of BRCA-positive Advanced Breast Cancer
Acronym: ICEBERG 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: KuDOS Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KU36-44; D0810C00008; 2006-006458-91 (EudraCT Number)
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Breast Neoplasms
Keywords: Advanced breast cancer; Poly(ADP ribose) polymerases; AZD2281,KU-0059436 (olaparib); BRCA1 protein; BRCA2 protein
MeSH Terms: conditions — Breast Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaparib 100 mg (Experimental): Participants will receive two 50 mg capsules in the morning and two 50 mg capsules in the evening in 28-days cycle until confirmed disease progression, continuous treatment interruption, unacceptable toxicity or any other discontinuation criterion is met.
  Interventions: Drug: Olaparib
- Olaparib 400 mg (Experimental): Participants will receive eight 50 mg capsules in the morning and eight 50 mg capsules in the evening in 28-days cycle until confirmed disease progression, continuous treatment interruption, unacceptable toxicity or any other discontinuation criterion is met.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Participants will receive capsules of olaparib orally as stated in arm description.
  Other Names: AZD2281; KU-0059436

SUMMARY:
The purpose of the study is to see if the drug KU-0059436 (olaparib) is effective and well tolerated in treating participants with measurable breast cancer gene (BRCA)1- or BRCA2-positive advanced breast cancer and for whom no curative therapeutic option exists.

DETAILED DESCRIPTION:
This is a Phase II, open-label, non-comparative, international, multicenter study to assess the efficacy and safety of olaparib when given orally twice daily (bd) in participants with advanced BRCA1- or BRCA2- associated breast cancer. Two sequential participant cohorts will receive continuous oral olaparib in 28-day cycles. The first cohort will receive 400 mg bd and the second cohort will receive 100 mg bd.

ELIGIBILITY:
Inclusion Criteria:

* Advanced breast cancer with positive BRCA1 or BRCA2 status
* Failed at least one prior chemotherapy
* In investigators opinion, no curative standard therapy exists
* Measurable disease

Exclusion Criteria:

* Brain metastases
* Less than 28 days since last treatment used to treat the disease
* Considered a poor medical risk due to a serious uncontrolled disorder

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-06-15 (Actual); Primary Completion 2009-02-27 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Carmichael, BSc, MBChB, MD, FRCP, Study Director — KuDOS Pharmaceuticals Limited; Andrew Tutt, PhD MRCP FRCR, Principal Investigator — Guy's and St Thomas's NHS Foundation Trust, London, UK
Locations (17):
- United States (2):
  - Research Site, West Hollywood, California
  - Research Site, Boston, Massachusetts
- Australia (2):
  - Research Site, Melbourne
  - Research Site, Randwick
- Research Site, Duarte, CA, Canada
- Germany (3):
  - Research Site, Cologne
  - Research Site, Kiel
  - Research Site, München
- Research Site, Tel Aviv, Israel
- Spain (2):
  - Research Site, Hospitalet deLlobregat
  - Research Site, Madrid
- Research Site, Lund, Sweden
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Edinburgh
  - Research Site, Fulham
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Tutt A, Robson M, Garber JE, Domchek SM, Audeh MW, Weitzel JN, Friedlander M, Arun B, Loman N, Schmutzler RK, Wardley A, Mitchell G, Earl H, Wickens M, Carmichael J. Oral poly(ADP-ribose) polymerase inhibitor olaparib in patients with BRCA1 or BRCA2 mutations and advanced breast cancer: a proof-of-concept trial. Lancet. 2010 Jul 24;376(9737):235-44. doi: 10.1016/S0140-6736(10)60892-6. Epub 2010 Jul 6. PMID 20609467

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 centers in 5 countries (Australia, Germany, Sweden, UK and the USA).
Pre-assignment Details: A total of 54 participants were enrolled in this study.
Groups:
- Olaparib 100 mg: Participants received two 50 mg capsules in the morning and two 50 mg capsules in the evening in 28-days cycle until confirmed disease progression, continuous treatment interruption, unacceptable toxicity or any other discontinuation criterion was met.
- Olaparib 400 mg: Participants received eight 50 mg capsules in the morning and eight 50 mg capsules in the evening in 28-days cycle until confirmed disease progression, continuous treatment interruption, unacceptable toxicity or any other discontinuation criterion was met.
Period: Overall Study
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Started | 27 | 27
Completed | 13 | 18
Not Completed | 14 | 9
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease progression | 11 | 8
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set comprised of all enrolled participants with positive BRCA status, who took at least one dose of investigational medicinal product irrespective of whether they completed the trial schedule and IMP regime or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 100 mg | Olaparib 400 mg | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (11.99) | 44.7 (9.55) | 44.7 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 21 | 19 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 25 | 26 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: The ORR is the percentage of participants whose best tumor response is either complete response (CR) or partial response (PR), according to the RECIST v1.0 criteria. The CR is defined as disappearance of all target lesions (TLs). The PR is defined as at least a 30% decrease in the sum of longest diameters (LD) taking as reference the baseline sum of LD. Percentage of participants with ORR is reported.
Time Frame: Baseline (Days -28 to 0), Day 1 of Cycle 3, thereafter every alternate cycles until study termination or withdrawal (approximately up to 2 years)
Population: The per-protocol (PP) population included all enrolled participants who completed the trial schedule and medication regime without any major deviations to the protocol.
Measure: Number; unit: Percentage of participants
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Number analyzed (Participants) | 24 | 26
Percentage of participants | 25.0 | 42.3

2. Secondary Outcome: Duration of Response (DoR) to Olaparib
Description: Duration of response is defined as the date of progression per RECIST criteria - the date when CR or PR [whichever is earliest] is confirmed + 1. The CR is defined as disappearance of all TLs. The PR is defined as at least a 30% decrease in the sum of LD taking as reference the baseline sum of LD. Duration of response was analyzed for those participants who had OR.
Time Frame: as for outcome 1
Population: The PP population included all enrolled participants who completed the trial schedule and medication regime without any major deviations to the protocol.
Measure: Median (Full Range); unit: Days
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Number analyzed (Participants) | 6 | 11
Days | 140.5 (55) [55 to 175] | 144.0 (92) [92 to 393]

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The CBR is defined as the percentage of participants with a RECIST tumor response of confirmed CR, PR or stable disease (SD) for ≥ 8 weeks +/- 1 week visit window. The CR is defined as disappearance of all TLs. The PR is defined as at least a 30% decrease in the sum of LD taking as reference the baseline sum of LD. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum of LD since the treatment started.
Time Frame: From Day 1 of Cycle 3 through study withdrawal (approximately up to 2 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Number analyzed (Participants) | 24 | 26
Percentage of Participants | 70.8 (50.8) [50.8 to 85.1] | 84.6 (66.5) [66.5 to 93.9]

4. Secondary Outcome: Best Percentage Change in Tumor Size
Description: The tumor size is defined as the sum of the longest diameters as measured among all target lesions. At each assessment, the percentage change in tumor size is defined as 100 × 1 - (sum of all target lesion diameters at visit/sum of all target lesion diameters at baseline).
Time Frame: Baseline (Days -28 to 0) through study withdrawal (approximately up to 2 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Best percentage change in tumor size
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Number analyzed (Participants) | 24 | 26
Best percentage change in tumor size | -10.14 [-68.9 to 286.7] | -29.43 [-100.0 to 26.7]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from first dose to the earlier date of radiologic progression (as per RECIST criteria) or death by any cause in the absence of objective progression. Those participants who were withdrawn from the study without disease progression were regarded as censored at their last evaluable RECIST assessment. Where participants had not progressed at the termination of the study, they were also regarded as censored at their last evaluable RECIST assessment. PFS was analyzed using Kaplan-Meier estimate.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Number analyzed (Participants) | 24 | 26
Days | 122 [67 to 167] | 193.5 [140 to 226]

6. Secondary Outcome: Number of Participants With Improvement in Eastern Co-operative Oncology Group (ECOG) Performance Status Total Score From Baseline
Description: ECOG performance status is used by researchers to assess how a participant's disease is progressing. The scores are: 0=Fully Active, able to carry out work without restrictions; 1=Restricted activity and able to carry out light work or sedentary nature; 2=capable of self-care but unable to carry out work activities; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely Disabled, and totally confined to bed or chair; 5=Dead. Change in ECOG performance status was defined as improved (less than the baseline value), no change (same as at baseline), worsened (greater than the baseline value) or missing (score is missing or was not recorded at baseline). If no measurement was recorded at Cycle 1 Day 1, the change was calculated in relation to the last recorded ECOG value prior to Day 1.
Time Frame: Screening (Days -7 to 0), Day 1 Cycle 7 (ie, after completing 6 cycles of treatment) and study withdrawal (approximately up to 2 years).
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Number analyzed (Participants) | 27 | 27
Participants
  Cycle 7 Day 1: number analyzed (Participants) | 11 | 15
  Cycle 7 Day 1 | 1 | 6
  Withdrawal visit: number analyzed (Participants) | 14 | 22
  Withdrawal visit | 0 | 2

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 480 (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Number analyzed (Participants) | 27 | 27
Participants
  Any TEAE | 27 | 27
  Any TESAE | 5 | 9

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs From Baseline
Description: Number of participants with clinically significant changes in vital signs are reported. Vital sign parameters included body temperature, blood pressure, and pulse rate.
Time Frame: Day 1 through Day 480 (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Number analyzed (Participants) | 27 | 27
Participants
  Tachycardia | 1 | 0
  Supraventricular arrhythmia | 1 | 0

9. Secondary Outcome: Number of Participants With at Least 2-Grade Change From Baseline to Worst Toxicity Grade in Clinical Laboratory Parameters
Description: Number of participants with at least 2-grade change from baseline to worst toxicity grade in clinical laboratory parameters are reported. Laboratory parameters included hematology, clinical chemistry, and urinalysis.
Time Frame: Day 1 through Day 480 (maximum observed duration)
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
Number analyzed (Participants) | 27 | 27
Participants
  Hemoglobin | 2 | 3
  White blood cells | 5 | 11
  Absolute neutrophil count | 3 | 6
  Lymphocytes | 3 | 2
  Platelets | 0 | 2
  Activated partial thromboplastin time | 1 | 2
  Alanine aminotransferase | 2 | 3
  Aspartate aminotransferase | 3 | 1
  Alkaline phosphatase | 1 | 0
  Gamma glutamyl transferase | 4 | 2
  Albumin | 1 | 0
  Total bilirubin | 0 | 4
  Sodium (decrease) | 1 | 0
  Potassium (increase) | 0 | 1
  Creatinine | 0 | 2
  Glucose (increase) | 2 | 2
  Glucose (decrease) | 3 | 3
  Calcium (decrease) | 3 | 3
  Amylase | 1 | 0
  Lipase | 2 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to 480 (maximum observed duration)
Description: Safety population included all participants who received at least one dose of study drug.
Arm/Group | Olaparib 100 mg | Olaparib 400 mg
All-Cause Mortality (participants affected / at risk) | 3/27 | 6/27
Serious Adverse Events (participants affected / at risk) | 5/27 | 9/27
Other Adverse Events (participants affected / at risk) | 27/27 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 100 mg (N=27) | Olaparib 400 mg (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 100 mg (N=27) | Olaparib 400 mg (N=27)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (19) | 14 (17)
Vomiting (Gastrointestinal disorders) | 6 (8) | 10 (16)
Constipation (Gastrointestinal disorders) | 8 (8) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 8 (10)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 5 (5)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (3)
Fatigue (General disorders) | 17 (19) | 19 (25)
Oedema peripheral (General disorders) | 4 (4) | 6 (6)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Chest pain (General disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Oral candidiasis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (4)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Weight increased (Investigations) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 6 (9) | 10 (23)
Migraine (Nervous system disorders) | 1 (1) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (7) | 2 (2)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The plasma concentration data was analysed using a population approach and polyadenosine 5' diphosphoribose polymerase (PARP) inhibition data had already been obtained from Study D0810C00002. Hence no pharmacokinetic and PARP inhibition data are included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.